CLINICAL TRIAL: NCT00273182
Title: InSync Model 8040 (InSync) and InSync III Model 8042 (InSync III) Systems for Cardiac Resynchronization Therapy (CRT) - InSync Registry
Brief Title: InSync Model 8040 (InSync) and InSync III Model 8042 (InSync III) Registry
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: 187
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Results first posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-07

CONDITIONS: Heart Failure; Cardiomyopathy
Keywords: Heart Failure; Cardiomyopathy; Cardiac pacing; Cardiac resynchronization therapy
MeSH Terms: conditions — Heart Failure; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: Patients implanted with InSync Model 8040, InSync III Model 8042 , or Medtronic CRT-D system. A total of 1999 subjects were enrolled in the study. Of them, 1738 had successful post market implants of InSync Model 8040 (601 subjects), InSync III Model 8042 (512 subjects) and CRT-D devices (625 subjects). The rest 262 subjects came from two pre-market studies: the MIRACLE study added 141 subjects to InSync Model 8040, and the InSync III study added 121 subjects to the InSync III Model 8042. A total of 1014 subjects completed the study through 36 month follow up. Follow-up of 1000 subjects was required by the FDA to satisfy the conditions of approval.
  Interventions: Device: InSync Model 8040; Device: InSync III Model 8042

INTERVENTIONS:
Device: InSync Model 8040 — Subjects with sucessful implants of InSync Model 8040.
Device: InSync III Model 8042 — Subjects with successful implants of InSync III Model 8042

SUMMARY:
Heart failure is a progressive disease that decreases the pumping action of the heart. This may cause a backup of fluid in the heart and may result in heart beat changes.

When there are changes in the heart beat sometimes an implantable heart device is used to control the rate and rhythm of the heart beat. In certain heart failure cases, when the two lower chambers of the heart no longer beat in a coordinated manner, cardiac resynchronization therapy (CRT) may be prescribed. CRT is similar to a pacemaker. It is placed (implanted) under the skin of the upper chest. CRT is delivered as tiny electrical pulses to the right and left ventricles through three or four leads (soft insulated wires) that are inserted through the veins to the heart.

The purpose of this study is to monitor the long-term performance of the InSync Model 8040 (InSync) and InSync III Model 8042 (InSync III) systems for cardiac resynchronization therapy (CRT).

DETAILED DESCRIPTION:
Condition of Approval study for cardiac resynchronization therapy with pacemakers, and for the Attain left ventricular leads 2187, 2188, 4193, and 4194.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with an InSync Model 8040 or InSync III Model 8042, a right ventricular lead, and a Medtronic market-released left ventricular lead as part of a system to deliver cardiac resynchronization therapy.

Exclusion Criteria:

* Patients with a history of a previously failed placement of a currently investigational Medtronic left ventricular lead within 30 days of enrollment in the InSync Registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for use of a cardiac device
Sampling Method: Non-Probability Sample
Enrollment: 1999 (Actual)
Dates: Start 2002-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: InSync Registry Study Leader, Study Chair — Medtronic
Locations (82):
- United States (82):
  - Birmingham, Alabama
  - Peoria, Arizona
  - Fort Smith, Arkansas
  - Little Rock, Arkansas
  - Long Beach, California
  - Napa, California
  - Oxnard, California
  - San Diego, California
  - Yuba City, California
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Rockford, Illinois
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Overland Park, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Salisbury, Maryland
  - Silver Spring, Maryland
  - Boston, Massachusetts
  - Worchester, Massachusetts
  - Detroit, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Marquette, Michigan
  - Saginaw, Michigan
  - Duluth, Minnesota
  - Minneapolis, Minnesota
  - Hattiesburg, Mississippi
  - Tupelo, Mississippi
  - Columbia, Missouri
  - Kansas City, Missouri
  - Saint Joseph, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Lincoln, Nebraska
  - Newark, New Jersey
  - Manhasset, New York
  - New York, New York
  - Rochester, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - High Pointe, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Mayfield Heights, Ohio
  - Oklahoma City, Oklahoma
  - Doylestown, Pennsylvania
  - Erie, Pennsylvania
  - Philadelphia, Pennsylvania
  - York, Pennsylvania
  - Providence, Rhode Island
  - Greenville, South Carolina
  - Spartanburg, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Lubbock, Texas
  - Sherman, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Johnson WB, Abraham WT, Young JB, Wheelan K, Smith AL, Chang Y, Brinkman P; InSync Registry Investigators. Long-term performance of the attain model 4193 left ventricular lead. Pacing Clin Electrophysiol. 2009 Sep;32(9):1111-6. doi: 10.1111/j.1540-8159.2009.02451.x. PMID 19719485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The InSync Registry commenced subject enrollment on February 27, 2002. A total of 1999 subjects were enrolled in the study during the time period of February 2002 through February 2008. 1014 subjects completed the study through 36 month follow up. Follow-up of 1000 subjects was required by the FDA to satisfy the conditions of approval.
Pre-assignment Details: 1999 subjects were enrolled in the study. Of them 1738 had successful post market implants of InSync Model 8040 (n=601), InSync III Model 8042 (n=512) and CRT-D devices (n=625). The rest 262 subjects came from two pre-market studies: MIRACLE study added 141 subjects to InSync Model 8040, InSync III study added 121 to InSync III Model 8042.
Groups:
- All Subjects: Patients successfully implanted with InSync Model 8040 (including post-market new implants of InSync Model 8040 and pre-market implants from the MIRACLE study), InSync III Model 8042 (including post-market new implants of InSync III Model 8042 and pre-market implants from the InSync III study), and post-market Medtronic CRT-D devices.
Period: Overall Study
Arm/Group | All Subjects
Started | 1999
Completed | 1014
Not Completed | 985
Not completed — Death | 450
Not completed — Lost to Follow-up | 88
Not completed — Withdrawal by Subject | 257
Not completed — Device/System Explant | 154
Not completed — Site exit, system change, 36 m FU missed | 36

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: Patients implanted with InSync Model 8040 (including post-market new implants of InSync Model 8040 and pre-market implants from the MIRACLE study), InSync III Model 8042 (including post-market new implants of InSync III Model 8042 and pre-market implants from the InSync III study), and post-market Medtronic CRT-D devices.
Arm/Group | All Subjects
Number analyzed (Participants) | 1999
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 686
  >=65 years | 1313
Age Continuous [Mean (Standard Deviation); unit: years] | 67.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 728
  Male | 1271
Region of Enrollment [Number; unit: participants]
  United States | 1999

OUTCOME MEASURES:

1. Primary Outcome: Overall Death Rate and Cause Specific Death Rate During Three Years Post Implant.
Description: Survival curves of overall mortality and cause specific mortality (due to progressive heart failure and sudden cardiac death) were created based on Kaplan-Meier estimates. Estimates went out to 36 month time point. Confidence intervals were calculated on a log-log scale. The Kaplan-Meier estimates are reported in the statistical analysis modules
Time Frame: 36 month follow-up
Population: The analysis included data from all subjects enrolled in the InSync Registry study and successfully implanted with the InSync or InSync III system.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 1999
participants
  Overall Death | 450
  Cause Specific Death | 213
Statistical Analysis 1: Comparison: All Subjects; For overall mortality, the endpoint is the proportion of subjects alive during three years post-implant. Survival curves of overall mortality and cause-specific mortality were created based on Kaplan-Meier (product limit) estimates. Confidence intervals will be calculated on a log-log scale; Test type: Superiority or Other; Kaplan-Meier (product limit) estimates — No p values for the analysis; Survival curves of cause-specific mortality were created based on Kaplan-Meier (product limit) estimates; Overall survival rate at 36 month = 71.0, 95% CI 2-sided [68.6 to 73.2] — The estimate is the overall survival rate at 36 month. left-truncation methods were used in the survival analysis for previously implanted subjects
Statistical Analysis 2: Comparison: All Subjects; For cause-specific mortality, the endpoint is the proportion of patients who are alive or do not die due to the progressive heart failure or sudden cardiac death causes during 3 years post-implant. Survival curves of cause-specific mortality were created based on Kaplan-Meier (product limit) estimates. Confidence intervals were calculated on a log-log scale; Test type: Superiority or Other; Kaplan-Meier (product limit) estimates — No p value for this analysis; Cause specific survival rate at 36 month; Cause specific survival rate at 36 month = 85.3, 95% CI 2-sided [83.3 to 87.1] — left-truncation methods were used in the survival analysis for previously implanted subjects

2. Secondary Outcome: Left Ventricular (LV) Lead R-wave Amplitude
Description: Summary statistics such as mean and 95% CI for the LV lead R-wave amplitude during the 36 months of follow-up.
Time Frame: 36 month follow-up
Population: 1999 subjects successfully implanted with a left ventricular lead as part of a Medtronic CRT/CRT-D system.
Measure: Mean (95% Confidence Interval); unit: mV
Arm/Group | All Subjects
Number analyzed (Participants) | 1999
mV
  6 months follow-up | 13.7 [13.4 to 14.1]
  12 months follow-up | 13.3 [13.0 to 13.7]
  18 months follow-up | 13.2 [12.8 to 13.6]
  24 months follow-up | 13.2 [12.8 to 13.6]
  30 months follow-up | 13.4 [13.0 to 13.8]
  36 months follow-up | 13.6 [13.1 to 14.1]

3. Secondary Outcome: Left Ventricular (LV) Lead Impedance
Description: Summary statistics such as mean and 95% CI for the LV lead impedance during the 36 months of follow-up.
Time Frame: 36 months follow-up
Measure: Mean (95% Confidence Interval); unit: ohms
Arm/Group | All Subjects
Number analyzed (Participants) | 1999
ohms
  6 months follow-up | 620 [609 to 630]
  12 months follow-up | 625 [613 to 636]
  18 months follow-up | 628 [615 to 641]
  24 months follow-up | 622 [608 to 635]
  30 months follow-up | 632 [617 to 646]
  36 months follow-up | 633 [619 to 648]

4. Secondary Outcome: Left Ventricular (LV) Lead Pacing Voltage Threshold
Description: Summary statistics such as mean and 95% CI for the LV lead pacing voltage threshold during the 36 months of follow-up
Time Frame: 36 months follow-up
Measure: Mean (95% Confidence Interval); unit: Volts
Arm/Group | All Subjects
Number analyzed (Participants) | 1999
Volts
  6 months follow-up | 1.70 [1.63 to 1.77]
  12 months follow-up | 1.65 [1.59 to 1.72]
  18 months follow-up | 1.69 [1.62 to 1.77]
  24 months follow-up | 1.72 [1.64 to 1.81]
  30 months follow-up | 1.76 [1.67 to 1.85]
  36 months follow-up | 1.76 [1.67 to 1.85]

5. Secondary Outcome: Subjects With Left Ventricular (LV) Lead Related Complications During Three Years Post-implant
Description: A left ventricular lead related complication is defined as an adverse event that requires invasive intervention or leads to loss of significant device function resulting from the presence or performance of the LV lead.
  Kaplan-Meier method was used to estimate complication-free rate during the three years of follow-up. Time to the first post-implant LV lead related complication was used for the calculation. Confidence intervals were calculated on a log-log scale.
Time Frame: 36 months follow-up
Population: The analysis included data from all subjects enrolled in the InSync Registry study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 1999
participants | 176
Statistical Analysis 1: Comparison: All Subjects; Kaplan-Meier (product limit) estimate of the curve representing the time to first post-implant LV lead related complication were calculated to the first time point where fewer than 50 patients are still at risk. Confidence intervals will be calculated on a log-log scale; Test type: Superiority or Other; Kaplan-Meier (product limit) estimate — No p value for this analysis; event free rate = 89.8, 95% CI 2-sided [88.3 to 91.2]

ADVERSE EVENTS:
Time Frame: 36 months
Groups:
- All Patients: The analysis included data from all subjects enrolled in the InSync Registry study.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 450/1999
Other Adverse Events (participants affected / at risk) | 175/1999
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=1999)
Death (General disorders) | 450 (450) — Death and adverse events which resulted in hospitalization are listed as serious adverse events. There was no AE resulted in hospitalization in this study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=1999)
4194 lv lead explanted (General disorders) | 1 (1) — Only LV lead related AEs are reported for this study.
Elevated pacing thresholds (General disorders) | 18 (18)
Exit block (General disorders) | 1 (1)
Failure to capture, loss of capture (General disorders) | 40 (41)
Heart failure decompensation (General disorders) | 1 (1)
Hypotension (General disorders) | 1 (1)
Lead conductor fracture (General disorders) | 2 (2)
Lead dislodgment (General disorders) | 70 (75)
Lead insulation failure (General disorders) | 1 (1)
Muscle stimulation-diaphragm (General disorders) | 47 (49)
Other (IPG code) (General disorders) | 1 (1)
Oversensing (General disorders) | 1 (1)
Pacemaker mediated tachycardia (General disorders) | 1 (1)
Pocket erosion (General disorders) | 1 (1)
Suboptimal position of 4194 lead (General disorders) | 1 (1)
Unable to defibrillate (General disorders) | 1 (1)
Undersensing (General disorders) | 2 (2)
Ventricular fibrillation (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators ("PI") to publish per the publication strategy/Clinical Investigation Plan following Medtronic's review for (a) disclosure of confidential information ("CI"), and (b) selection and order of publications by the publications committee. Any such CI is deleted prior to publication/presentation. Medtronic may not otherwise censor/interfere with the publication. PI's may not publish single-site data until the main multi-site publication has occurred.